CLINICAL TRIAL: NCT05148702
Title: The EXTEND Trial: Fixed-extended-duration Antibiotics (28 Days) Compared to Standard Care Antibiotic Durations in Adult Patients With Complicated Intra-abdominal Infection and Their Impact on Treatment Failure
Brief Title: EXTENDed Antibiotic Durations Compared to Standard Durations for Patients With Complicated Intra-abdominal Infection.
Acronym: EXTEND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarah Cockayne (Other)
Collaborators: University of York (Other); University of Birmingham (Other); Chesterfield Royal Hospital NHS Foundation Trust (Unknown); University of Leeds (Other); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor-Investigator, Sarah Cockayne, Research Fellow, University of York
Organization: University of York (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIHR131784; ISRCTN 72819021 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2021-11-19; First posted 2021-12-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Complicated Intra-abdominal Infection
Keywords: infection; antibiotics; antibiotic resistance
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: A phase III multicentre, open label, two-arm, parallel group, pragmatic, randomised controlled trial with internal pilot.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Clinician decided antibiotic treatment duration
  Interventions: Drug: Antibiotic - standard duration
- Fixed-extended-duration antibiotics (Experimental): 28 day antibiotic treatment duration
  Interventions: Drug: Antibiotic - fixed-extended-duration

INTERVENTIONS:
Drug: Antibiotic - standard duration — Clinician decided antibiotic and duration of treatment
  Arms: Standard care
Drug: Antibiotic - fixed-extended-duration — Clinician decided antibiotic for a fixed duration of 28 days.
  Arms: Fixed-extended-duration antibiotics

SUMMARY:
A multicentre, open label, two-arm, parallel group, pragmatic, randomised controlled trial with internal pilot. A total of 1166 consenting adult patients with cIAI will be recruited and randomised on a 1:1 basis between 28-days antibiotics and standard care antibiotics. Patients will be followed up for 180 days to determine cost effectiveness and the rate of treatment failure in each group.

DETAILED DESCRIPTION:
UK data suggests that current treatment for complicated intra-abdominal infections (cIAIs) results in unacceptably high rates of cIAI relapse and extra-abdominal infection. As a guiding rule, shorter antibiotic durations are important to combat antimicrobial resistance, but this is not true when these shorter courses need repeating and result in more days in hospital. Optimal care for patients should be our primary concern.

The EXTEND trial aims to find out whether a fixed extended duration of 28 days of antibiotics is superior to the current standard duration (typically 7-18 days) based on clinical outcomes and quality of life assessed over 180 days of follow up. Cost effectiveness will also be determined.

A target of 1166 patients will be recruited from ICUs and hospital in-patient wards across approximately 30 NHS trust hospitals. Only patients that are able provide consent (or those with a consultee able to confirm whether the patient would wish to be included in the study) can take part in the trial. They will receive antibiotics as prescribed by their treating clinician, but the duration of treatment will be determined by randomisation. Patients will have equal chance of randomisation to the standard care arm, in which the antibiotic duration will be determined by the treating clinician, or the intervention arm, a fixed duration of 28 days treatment.

Patients (or a personal consultee) will complete a quality of life questionnaire at baseline and 30, 60 and 180 days after randomisation. At follow-up timepoints they will also complete questionnaires on antibiotic use and health care resource use. Hospital notes will be used to collect data on inpatient admissions, relapse and further infections.

The study is Sponsored by the University of Leeds

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 16 years) with cIAI* (see cIAI definition)
* Being treated with antibiotics until the point of randomisation, but within 10 days of initiation of effective antibiotic treatment** for cIAI
* Ability to provide informed consent by the patient or their consultee.
* More than 72 hours*** of active in-patient management for the patients cIAI is required
* In the event that the patient is re-admitted to hospital during the trial period, they are likely to be admitted to a hospital participating in the EXTEND trial.

Patients will be included in the trial whether or not they undergo surgical or radiological source control procedures.

* cIAI is defined by the following case definition:

* A clinical presentation consistent with cIAI, plus
* Fever (temperature of ≥ 37.8°C) and/or a neutrophilia (> 7.5×109/L) and/or neutropaenia (<1.8 x 109 /L) and/or intestinal pathogens cultured from sterile sites (closed peritoneum or blood) around the time of cIAI diagnosis, plus
* Evidence of pathologic findings on radiologic examination, or
* Evidence of pathologic findings at operation

  ** The first day of effective antibiotic treatment will be determined by the patient's clinical team or clinical research team. Antibiotics that do not count towards these 10 days of effective treatment are:
* Antibiotic prophylaxis e.g., penicillin for splenectomy, elective surgery antibiotic prophylaxis, UTI prophylaxis
* Treatment for other infections that is not effective for cIAI e.g., cystitis. Antibiotics that re often used for cystitis and aren't effective for cIAI include Cephalexin, Fosfomycin Trimethoprim, Nitrofurantoin, and Pivmecillinam.
* Oral antibiotics prescribed to treat infection prior to hospitalisation
* Previous courses of treatment antibiotics: A previous course is one stopped for 48 hours or more

  * The further 72 hours starts from the first day of effective antibiotic treatment i.e., for a patient admitted to hospital with a cIAI, 3 days of admission are needed. Where a patient is already in hospital e.g., a post operative patient, a further 3 days of admission are required starting from the point of the first day of effective antibiotic treatment.

Exclusion Criteria:

* Perforated gastric ulcer or duodenal ulcer treated within 24 hours of the onset of symptoms.
* Traumatic injury to the bowel (including iatrogenic or intra-operative) treated within 12 hours of injury.
* Uncomplicated diverticulitis defined as an episode with a short history and with clinical signs of diverticulitis, with an increased body temperature and inflammatory parameters, verified by computed tomography (CT), and without any sign of complications such as abscess, free air or fistula.
* Grade 1 to 3 appendicitis. To be eligible patient must have Grade 4 or 5 appendicitis defined by the 2017 American Association for the Surgery Trauma Grading System with either generalised peritonitis at surgery, or no or partial source control e.g. radiological drainage
* Non-perforated cholecystitis.
* Ischemic or necrotic intestine without perforation
* Uterine perforation following uterine surgery treated <six hours following injury.
* cIAIs with a low risk of complications who may receive more than 72 hours antibiotics are not intended to be included, such as those listed above. Traumatic injury to the bowel (including iatrogenic or intra-operative) treated within 12 hours of injury, Uterine perforation following uterine surgery treated within six hours of injury, Perforated gastric ulcer or duodenal ulcer treated within 24 hours of the onset of symptoms). Clinician assessment on the eligibility of patients receiving more than 72 hours of in-patient surgical care and antibiotics for their cIAI may be required in patients who have clinically improved at this point and do not require active surgical care but remain in hospital and on antibiotics.
* Current enrolment in another trial dictating antibiotic treatment duration.
* Previous Clostridium difficile infection
* Infected necrotic pancreatitis
* Concomitant infection requiring ≥4 weeks antibiotic therapy including Intra-hepatic abscess/es planned to be treated with fixed-extended-duration antibiotics of 4 to 6 weeks antibiotics, osteomyelitis, and endocarditis.
* Peritoneal dialysis
* Previously recruited for the EXTEND trial
* Treatment with Interleukin-6 Inhibitors
* High likelihood of death within 72 hours of cIAI randomisation in the opinion of the local Investigator
* Limitations in treatment decided before inclusion. Limitations in treatment that exclude patients from the EXTEND trial are those clinical decisions linked to an expectation the patient will die during this episode of infection.
* Patient with persistent cIAI of more than 6 months duration

A maximum of 20% of participants entering the trial can have a source of cIAI as the appendix. If 230 patients with appendix as the source are recruited, this will become an exclusion criteria for subsequent patients.

Note: There are absolute exclusions that preclude trial participation. These include: C. difficile infection, Infected necrotic pancreatitis, Concomitant infection requiring ≥4 weeks antibiotic therapy, Treatment with Interleukin-6 Inhibitors, High likelihood of death within 72 hours of randomisation, Limitations in treatment decided before inclusion, Peritoneal dialysis, Previously recruited for the EXTEND trial, Patient with persistent cIAI of more than 6 months duration and a patient with persistent cIAI of more than 6 months duration. If a patient has two intraabdominal infections, the presence of one of the following ineligible infections does not make a patient ineligible if the other cIAI is eligible: Perforated gastric ulcer or duodenal ulcer treated within 24 hours of the onset of symptoms, Traumatic injury to the bowel (including iatrogenic or intra-operative) treated within 12 hours of injury, Uncomplicated diverticulitis, Ineligible cases of appendicitis (see exclusion criteria above), Uncomplicated cholecystitis, Ischemic or necrotic intestine without perforation, Uterine perforation following uterine surgery treated within six hours of injury or cIAI with a low risk of complications.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1166 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure within 180 days of randomisation. | 180 days
  For in-patients, treatment failure is defined when a patient meets objective criteria for both inflammation and infection within a 5 day period. Meeting of the criteria for inflammation may precede or follow the date that criteria for infection were met (the first day of an eligible antibiotic treatment course). These criteria are:
  Criteria for Inflammation
  * A fever (≥ 37.8 degrees Celsius) or hypothermia (≤36 degrees Celsius), plus
  * A neutrophilia (>7.5 x109/L) or neutropaenia (<1.8 x 109/L), plus
  * A CRP over 100 mg/L
  PLUS, criteria for infection
  * Initiation of a new antibiotic treatment course of ≥ 5 days, or
  * A change in antibiotic treatment continued for ≥ 5 days, or
  * Initiation of a new antibiotic treatment, or a change in antibiotic treatment, and death within 5 days.
  * Bacteraemia with a recognised intestinal pathogen include: Anaerobes (e.g., Bacteroides), Enterobacterales and Streptococcus species.
  Assessed by blinded outcome committee

SECONDARY OUTCOMES:
Quality of life (EQ-5D-5L) | 180 days
  Participants will complete the EQ-5D-5L at baseline, and at 30, 90 and 180 days post-randomisation.
Cost effectiveness | 180 days
  Participants will complete health care resource use questionnaires at 30, 90 and 180 days after randomisation to record activity outside of hospital. Research teams will record data related to expenses as an inpatient.
Desirability Of Outcome Ranking (DOOR) | 180 days
  Patients will be categorised according to the worst outcome they experience over the 6 months follow up period using a four-level ordinal classification the Desirability Of Outcome Ranking (DOOR). The four levels will be C1 = No treatment failure, C2 = Treatment failure (as for the primary outcome), C3 = Treatment failure associated with sepsis (NEWS 6 in ward-based patients and SOFA 2 in ICU based patients) and C4 = Treatment failure associated with death.
Number and type of source control procedures | 180 days
  The total number and type of source control procedures measured by reviewing patient notes at 180 days after randomisation. The definition of source control used for this study is any procedure that stops the ongoing contamination of the peritoneal cavity and removes the majority of the contaminated intraperitoneal contents to the extent that no further acute interventions are felt to be necessary.
  The different types (radiological, surgical) and source control procedures of any type occurring in each randomised group will be compared using a proportional odds model, with fixed effects for allocation, the stratification factors and other prognostic baseline covariates, and random intercepts for study recruitment site.
Relapse of cIAI | 180 days
  The proportion of patients that experience a relapse of cIAI during the 180 days following randomisation will be reported by randomised group.
All-cause mortality | 180 days
  All-cause mortality (time to event) measured by reviewing patient notes at 180 days after randomisation.
  Brief summaries of the total time at risk and number/proportion of participants who died will be presented by randomised group and overall
Length of hospital stay | 180 days
  Length of hospital stay measured by reviewing patient notes at 180 days after randomisation. Total number of nights in hospital (with death coded as the worst/highest outcome) will be compared using a proportional odds model, with fixed effects for allocation, the stratification factors and other prognostic baseline covariates, and random intercepts for study recruitment site.
Re-admission | 180 days
  Re-admission measured by reviewing patient notes at 180 days after randomisation.
  The proportion of participants who are re-admitted to hospital during the 180 days following randomisation, and number of re-admissions per participant will be reported descriptively by randomised group and overall
C. difficile infection | 180 days
  C. difficile infection measured by reviewing patient notes at 180 days after randomisation.
  The proportion of patients that experience C. difficile infection during the 180 days following randomisation will be reported by randomised group.
Anti-microbial resistant (AMR) infections | 180 days
  Anti-microbial resistant (AMR) infections measured by reviewing patient notes at 180 days after randomisation. When standard treatment fails in patients with cIAI, antibiotics are often escalated to one of the carbapenem class of antibiotics. We will therefore use rates of carbapenem prescribing as a surrogate for AMR infections.
  Participants will undergo passive surveillance for antimicrobial resistant infections (including MRSA, VRE, ESBL and CPE) during the 180 days following randomisation. The proportion of patients that experience each type of antimicrobial infection, number of days receiving carbapenem class antibiotics and the number of antibiotic class switches will be reported descriptively by randomised group and overall.
Days of antibiotic therapy (in-patient and outpatient) | 180 days
  Days of antibiotic therapy (in-patient and outpatient) including anti-fungal therapy measured by reviewing patient notes and from a questionnaire completed by patients at 180 days after randomisation.
  The total number of days of anti-microbial therapy (inpatient, outpatient and overall) during the 180 days following randomisation, proportion of total follow up time on anti-microbial therapy, and mortality will be reported descriptively by randomised group and overall.
Acute kidney injury | 180 days
  Acute kidney injury measured by reviewing patient notes at 180 days after randomisation and defined as: an increase in serum creatinine by ≥ 0.3 mg/dl (≥ 26.5 µmol/l) within 48 hours; or increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or urine volume < 0.5 ml/kg/h for 6 hours (KDIGO Clinical Practice Guideline for Acute Kidney Injury).
  The proportion of patients that experience acute kidney injury during the 180 days following randomisation will be reported by randomised group.
Complications | 180 days
  Will be measure by reviewing patient notes at 180 days after randomisation.
Number of days on ventilation and days of renal replacement therapy. | 180 days
  Will be measure by reviewing patient notes at 180 days after randomisation.
Time to treatment failure | 180 days.
  Time to treatment failure and number of episodes of treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kirby, MD, Principal Investigator — University of Leeds
Locations (36):
- United Kingdom (36):
  - Cwm Taf Morgannwg University Health Board,, Abercynon
  - NHS Grampian, Aberdeen
  - Hywel Dda University Health Board, Aberystwyth
  - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - UniversityHospitals Birmingham NHS Foundation Trust, Birmingham
  - Bolton NHS Foundation Trust, Bolton
  - United Lincolnshire Hospitals NHS Trust - Pilgrim Hospital Boston, Boston
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - North Bristol NHS Trust, Bristol
  - North Cumbria Integrated Care NHS Foundation Turst, Carlisle
  - Chesterfield Royal Hospital NHS Foundation Trust, Chesterfield
  - University Hospital Coventry & Warwickshire, Coventry
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - Northern Lincolnshire and Goole NHS Foundation Trust - Grimsby, Grimsby
  - Hull University Teaching Hospitals NHS Trust, Hull
  - East Suffolk and North Essex NHS Foundation Trust, Ipswich
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King'S College Hospital Nhs Foundation Trust, London
  - East Cheshire NHS Trust, Macclesfield
  - Manchester University NHS Foundation Trust, Manchester
  - Aneurin Bevan University Health Board, Newport
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospital NHS Trust, Nottingham
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Barking, Havering and Redbridge University Hospitals Nhs Trust, Romford
  - East Sussex Hospitals NHS Trust, Saint Leonards-on-Sea
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Royal Cornwall Hospitals NHS Trust, Truro
  - University Hospitals Sussex NHS Foundation Trust, Worthing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial website — https://www.york.ac.uk/healthsciences/research/trials/ytutrialsandstudies/trials/extend/